CLINICAL TRIAL: NCT00293254
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Antiretroviral Activity of MK-0518 in Combination With an Optimized Background Therapy (OBT), Versus Optimized Background Therapy Alone, in HIV-Infected Patients With Documented Resistance to at Least 1 Drug in Each of the 3 Classes of Licensed Oral Antiretroviral Therapies
Brief Title: A Study to Evaluate the Safety and Efficacy of Raltegravir (MK0518) in HIV-Infected Patients Failing Current Antiretroviral Therapies (0518-019)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0518-019; 2005_097
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2009-09-30 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): raltegravir potassium
  Interventions: Drug: raltegravir potassium
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: raltegravir potassium — Raltegravir 400 mg twice daily (b.i.d.) by mouth (p.o.) with optimized background therapy. Treatment period of 48 weeks.
  Other Names: ISENTRESS™
  Arms: 1
Drug: Comparator: placebo — Placebo p.o. b.i.d. with optimized background therapy. Treatment period of 48 weeks.
  Arms: 2

SUMMARY:
This study will investigate the safety and efficacy of raltegravir as a therapy for Human Immunodeficiency Virus (HIV)-infected patients failing current therapy with 3-class antiviral resistance.

DETAILED DESCRIPTION:
The primary double-blind study of raltegravir versus placebo was extended to 156 weeks and was followed by an open-label raltegravir phase in which continuing participants from both the raltegravir and placebo groups received open-label raltegravir for an additional 84 weeks for a maximum duration of up to 240 weeks. Participants who had viral failure after Week 16 may have received open-label raltegravir until Week 240.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be HIV positive with HIV RNA values that are within ranges required by the study
* Patient must have documented failure of certain antiretroviral therapy
* Patient must be on the same antiretroviral therapy for at least the past two months

Exclusion Criteria:

* Patient less than 16 years old
* Additional study criteria will be discussed and identified by the study doctor

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Steigbigel RT, Cooper DA, Kumar PN, Eron JE, Schechter M, Markowitz M, Loutfy MR, Lennox JL, Gatell JM, Rockstroh JK, Katlama C, Yeni P, Lazzarin A, Clotet B, Zhao J, Chen J, Ryan DM, Rhodes RR, Killar JA, Gilde LR, Strohmaier KM, Meibohm AR, Miller MD, Hazuda DJ, Nessly ML, DiNubile MJ, Isaacs RD, Nguyen BY, Teppler H; BENCHMRK Study Teams. Raltegravir with optimized background therapy for resistant HIV-1 infection. N Engl J Med. 2008 Jul 24;359(4):339-54. doi: 10.1056/NEJMoa0708975. PMID 18650512
- [Background] Cooper DA, Steigbigel RT, Gatell JM, Rockstroh JK, Katlama C, Yeni P, Lazzarin A, Clotet B, Kumar PN, Eron JE, Schechter M, Markowitz M, Loutfy MR, Lennox JL, Zhao J, Chen J, Ryan DM, Rhodes RR, Killar JA, Gilde LR, Strohmaier KM, Meibohm AR, Miller MD, Hazuda DJ, Nessly ML, DiNubile MJ, Isaacs RD, Teppler H, Nguyen BY; BENCHMRK Study Teams. Subgroup and resistance analyses of raltegravir for resistant HIV-1 infection. N Engl J Med. 2008 Jul 24;359(4):355-65. doi: 10.1056/NEJMoa0708978. PMID 18650513
- [Result] Steigbigel RT, Cooper DA, Teppler H, Eron JJ, Gatell JM, Kumar PN, Rockstroh JK, Schechter M, Katlama C, Markowitz M, Yeni P, Loutfy MR, Lazzarin A, Lennox JL, Clotet B, Zhao J, Wan H, Rhodes RR, Strohmaier KM, Barnard RJ, Isaacs RD, Nguyen BY; BENCHMRK Study Teamsa. Long-term efficacy and safety of Raltegravir combined with optimized background therapy in treatment-experienced patients with drug-resistant HIV infection: week 96 results of the BENCHMRK 1 and 2 Phase III trials. Clin Infect Dis. 2010 Feb 15;50(4):605-12. doi: 10.1086/650002. PMID 20085491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 3; First Patient In: 08-Mar-2006; Last Patient Last Visit (LPLV) for Week 48: 31-Jul-2007; Extension Study LPLV Week 240: May 2011
  53 sites (US, Brazil, Canada, Colombia, Mexico, and Puerto Rico).
Pre-assignment Details: Patients failed prior antiretroviral therapy (HIV RNA >1000 copies/mL), and had documented resistance to at least one drug in each class of licensed oral antiretroviral therapy (Nucleoside Reverse Transcriptase inhibitors, Non-Nucleoside Reverse Transcriptase Inhibitors, and Protease Inhibitors). All patients must have met laboratory criteria.
Period: Primary Study - Double-Blind Week 0-48
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Started | 232 | 119
Treated | 230 | 119
Continuing in Double-Blind | 177 (Excludes participants who entered the Open-Label Post-Virologic Failure (OLPVF) Phase) | 55 (Excludes participants who entered the OLPVF phase)
Completed | 177 | 55
Not Completed | 55 | 64
Not completed — Never Treated | 2 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Death | 5 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Moved or trial terminated at site | 1 | 0
Not completed — Entered OLPVF Phase | 35 | 57
Period: Extension - Double-Blind Week 49-156
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Started | 177 | 54 (1 of 55 participants who completed Week 48 did not enter the extension study.)
Completed | 120 | 25
Not Completed | 57 | 29
Not completed — Adverse Event | 4 | 1
Not completed — Death | 4 | 1
Not completed — Lack of Efficacy | 3 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Participant Moved/Site Stopped Trial | 6 | 3
Not completed — Other Reason | 10 | 2
Not completed — Entered OLPVF Phase | 15 | 7
Period: Extension - Open-Label Week 157-240
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Started | 120 | 19 (6 of 25 participants who completed the double-blind phase did not enter this open-label phase.)
Completed | 110 | 18
Not Completed | 10 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other Reason | 4 | 0
Period: Open-Label Post Virologic Failure Phase
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Started | 50 (Number of participants who failed treatment and consented to enter the OLPVF phase) | 64 (Number of participants who failed treatment and consented to enter the OLPVF phase)
Completed | 19 | 37
Not Completed | 31 | 27
Not completed — Adverse Event | 4 | 7
Not completed — Lack of Efficacy | 16 | 14
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Participant Moved/Site Stopped Trial | 1 | 1
Not completed — Other Reason | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT | Total
Number analyzed (Participants) | 230 | 119 | 349
Age, Continuous [Mean (Full Range); unit: Years] | 45.3 [16 to 67] | 46.5 [17 to 70] | 45.7 [16 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 210 | 107 | 317
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 127 | 77 | 204
  Black | 47 | 21 | 68
  Asian | 2 | 1 | 3
  Hispanic | 47 | 18 | 65
  Native American | 1 | 0 | 1
  Other | 6 | 2 | 8
Cluster of Differentiation 4 (CD4) Cell Count [Mean (Full Range); unit: cells/mm^3] | 146 [1 to 757] | 163 [0 to 674] | 152 [0 to 757]
Plasma Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) [Geometric Mean (Full Range); unit: copies/mL] | 49159 [200 to 750000] | 47850 [200 to 750000] | 48709 [200 to 750000]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving HIV RNA <400 Copies/mL at Week 16
Description: Percentage of participants who achieved HIV RNA <400 copies/mL at Week 16
Time Frame: 16 Weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 229 | 119
Percentage of Participants | 77.3 [71.3 to 82.6] | 42.9 [33.8 to 52.3]

2. Primary Outcome: Percentage of Participants Achieving HIV RNA <400 Copies/mL at Week 48
Description: Percentage of participants who achieved HIV RNA <400 copies/mL at Week 48
Time Frame: 48 Weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 228 | 119
Percentage of Participants | 71.1 [64.7 to 76.8] | 37.8 [29.1 to 47.2]

3. Primary Outcome: Double-Blind Extension - Week 156: Percentage of Participants Achieving HIV RNA <400 Copies/mL
Description: Percentage of participants who achieved HIV RNA <400 copies/mL at Week 156
Time Frame: 156 Weeks
Population: The analysis population was based on a non-completer equals failure approach where missing values for participants who discontinued the study for any reason were considered treatment failures.
  Participants who experienced virologic failure after Week 16 are counted also as treatment failures for the subsequent virologic efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 229 | 119
Percentage of Participants | 50.2 [43.6 to 56.9] | 21.0 [14.1 to 29.4]

4. Primary Outcome: Open-Label Extension - Week 240: Percentage of Participants Achieving HIV RNA <400 Copies/mL
Description: Percentage of participants who achieved HIV RNA <400 Copies/mL at Week 240
Time Frame: 240 Weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Raltegravir 400 mg b.i.d. + OBT: Raltegravir 400 mg b.i.d. plus OBT includes all participants initially randomized to raltegravir. Those who did not experience virologic failure by Week 156 may have continued into the open-label phase. During the open-label phase, these participants continued to receive raltegravir plus OBT until Week 240.
- Placebo + OBT: Placebo plus OBT includes all participants initially randomized to placebo. Those who did not experience virologic failure by Week 156 may have continued into the open-label phase. During the open-label phase, these participants received raltegravir plus OBT until Week 240.
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 230 | 119
Percentage of Participants | 45.7 [39.1 to 52.3] | 13.4 [7.9 to 20.9]

5. Secondary Outcome: Percentage of Participants Achieving HIV RNA <50 Copies/mL at Week 16
Description: Percentage of participants who achieved HIV RNA <50 copies/mL at Week 16
Time Frame: 16 Weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 229 | 119
Percentage of Participants | 62.0 [55.4 to 68.3] | 36.1 [27.5 to 45.4]

6. Secondary Outcome: Percentage of Participants Achieving HIV RNA <50 Copies/mL at Week 48
Description: Percentage of participants who achieved HIV RNA <50 copies/mL at Week 48
Time Frame: 48 Weeks
Population: Participants who experienced virologic failure after Week 16 are also counted as treatment failures for the subsequent virologic efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 228 | 119
Percentage of Participants | 59.6 [53.0 to 66.1] | 34.5 [26.0 to 43.7]

7. Secondary Outcome: Double-Blind Extension - Week 156: Percentage of Participants Achieving HIV RNA <50 Copies/mL
Description: Percentage of participants who achieved HIV RNA <50 copies/mL at Week 156
Time Frame: 156 Weeks
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 229 | 119
Percentage of Participants | 47.6 [41.0 to 54.3] | 17.6 [11.3 to 25.7]

8. Secondary Outcome: Open-Label Extension - Week 240: Percentage of Participants Achieving HIV RNA <50 Copies/mL
Description: Percentage of participants who achieved HIV RNA <50 copies/mL at Week 240
Time Frame: 240 Weeks
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 230 | 119
Percentage of Participants | 41.3 [34.9 to 48.0] | 13.4 [7.9 to 20.9]

9. Secondary Outcome: Double-Blind Extension - Week 156: Percentage of Participants Without Loss of Virologic Response
Description: For participants with confirmed HIV RNA levels <50 copies/mL on 2 consecutive visits, loss of virologic response is the occurrence of the first value >50 copies/mL or loss to follow-up; participants who never achieved HIV RNA <50 copies/mL on 2 consecutive visits are also considered as having loss of virologic response. Events are the numbers of participants with loss of virologic response versus the numbers of participants with no loss of virologic response (event-free).
Time Frame: 156 Weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 230 | 119
Percentage of Participants | 44.3 | 17.6

10. Secondary Outcome: Change From Baseline in HIV RNA (Log 10 Copies/mL) at Week 16
Description: Mean change from baseline at Week 16 in HIV RNA (log 10 copies/mL)
Time Frame: Baseline and Week 16
Population: Observed mean change from baseline in log10 plasma HIV RNA calculated using conventional imputation (replace <400 copies by 400 copies if signal detected; 200 copies if not detected); Missing values: Baseline carry-forward for all failures/discontinued due to lack of efficacy
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 222 | 117
HIV RNA (log10 copies/mL) | -1.92 [-2.05 to -1.78] | -1.06 [-1.26 to -0.86]

11. Secondary Outcome: Change From Baseline in HIV RNA (log10 Copies/mL) at Week 48
Description: Mean change from baseline at Week 48 in HIV RNA (log10 copies/mL)
Time Frame: Baseline and Week 48
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 216 | 114
HIV RNA (log10 copies/mL) | -1.75 [-1.90 to -1.59] | -0.87 [-1.08 to -0.67]

12. Secondary Outcome: Double-Blind Extension - Week 156: Change From Baseline in HIV RNA (log10 Copies/mL)
Description: Mean change from baseline at Week 156 in HIV RNA (log10 copies/mL)
Time Frame: Baseline and Week 156
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 189 | 102
HIV RNA (log10 copies/mL) | -1.37 [-1.55 to -1.20] | -0.52 [-0.71 to -0.33]

13. Secondary Outcome: Open-Label Extension - Week 240: Change From Baseline in HIV RNA (log10 Copies/mL)
Description: Mean change from baseline at Week 240 in HIV RNA (log10 copies/mL)
Time Frame: Baseline and Week 240
Population: Observed mean change from baseline in log10 plasma HIV RNA calculated using conventional imputation (replace <400 copies by 400 copies if signal detected; 200 copies if not detected); Missing values: Baseline carry-forward for all failures/discontinued due to lack of efficacy
  Participants with virologic failure after Week 16 = treatment failures
Measure: Mean (95% Confidence Interval); unit: HIV RNA (log10 copies/mL)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 182 | 95
HIV RNA (log10 copies/mL) | -1.31 [-1.49 to -1.13] | -0.41 [-0.59 to -0.23]

14. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at Week 16
Description: Mean change from baseline at Week 16 in CD4 cell count (cells/mm^3)
Time Frame: Baseline and Week 16
Population: Observed failure approach assuming baseline-carry-forward for all failures, exclude other missing values. Baseline CD4 cell count (cells/mm^3) was carried forward for participants who discontinued assigned therapy due to lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 219 | 117
CD4 Cell Count (cells/mm^3) | 85.8 [72.7 to 99.0] | 39.9 [26.2 to 53.6]

15. Secondary Outcome: Change From Baseline in CD4 Cell Count (Cells/mm^3) at Week 48
Description: Mean change from baseline at Week 48 in CD4 cell count (cells/mm^3)
Time Frame: Baseline and Week 48
Population: Observed failure approach assuming baseline-carry-forward for all failures, exclude other missing values. Baseline CD4 cell count (cells/mm^3) was carried forward for participants who discontinued assigned therapy due to lack of efficacy.
  Participants with virologic failure after Week 16 are treatment failures for virologic efficacy analyses.
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 217 | 114
CD4 Cell Count (cells/mm^3) | 98.4 [84.1 to 112.7] | 39.8 [23.5 to 56.1]

16. Secondary Outcome: Double-Blind Extension - Week 156: Change From Baseline in CD4 Cell Count(Cells/mm^3)
Description: Mean change from baseline at Week 156 in CD4 cell count (cells/mm^3)
Time Frame: Baseline and Week 156
Population: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm^3)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 189 | 101
CD4 Cell Count (cells/mm^3) | 157.2 [130.7 to 183.6] | 54.2 [30.0 to 78.3]

17. Secondary Outcome: Open-Label Extension - Week 240: Change From Baseline in CD4 Cell Count (Cells/mm^3)
Description: Mean change from baseline at Week 240 in CD4 cell count (cells/mm^3)
Time Frame: Baseline and Week 240
Population: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (Cells/mm^3)
Arm/Group | Raltegravir 400 mg b.i.d. + OBT | Placebo + OBT
Number analyzed (Participants) | 181 | 95
CD4 Cell Count (Cells/mm^3) | 172.1 [141.7 to 202.5] | 54.1 [27.1 to 81.0]

ADVERSE EVENTS:
Time Frame: 240 Weeks
Description: Adverse events are reported by original treatment group for the entire 240-week study, including double-blind, open-label, and OLPVF phases; 83 of 119 participants in the placebo group also received raltegravir in the open-label or OLPVF phase.
Groups:
- Raltegravir 400 mg b.i.d. Plus OBT: Includes all participants initially randomized to raltegravir, including those without virologic failure who
  continued into the open-label phase at Week 156 and those who entered the OLPVF phase due to virologic failure. During either open-label phase up to Week 240, these participants continued to receive raltegravir 400 mg b.i.d. plus OBT.
- Placebo Plus OBT: Includes all participants initially randomized to placebo, including those without virologic failure who continued into the open-label phase at Week 156 and those who entered the OLPVF phase due to virologic failure. During either open-label phase up to Week 240, these participants continued to receive raltegravir 400 mg b.i.d. plus OBT.
Arm/Group | Raltegravir 400 mg b.i.d. Plus OBT | Placebo Plus OBT
Serious Adverse Events (participants affected / at risk) | 80/230 | 54/119
Other Adverse Events (participants affected / at risk) | 214/230 | 111/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir 400 mg b.i.d. Plus OBT (N=230) | Placebo Plus OBT (N=119)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 1 (1)
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Blindness cortical (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Ileitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (2)
Death (General disorders) | 2 (2) | 3 (3)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Immune reconstitution syndrome (Immune system disorders) | 2 (2) | 1 (1)
AIDS dementia complex (Infections and infestations) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess bacterial (Infections and infestations) | 2 (3) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Acute HIV infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 3 (3)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Atypical mycobacterial lymphadenitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cryptococcosis (Infections and infestations) | 1 (1) | 0 (0)
Cryptosporidiosis infection (Infections and infestations) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 (1) | 3 (3)
Cytomegalovirus colitis (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (3)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1)
HIV wasting syndrome (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 2 (2) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 12 (17) | 5 (5)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 2 (2) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (4) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 2 (5)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kaposi's sarcoma AIDS related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 3 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir 400 mg b.i.d. Plus OBT (N=230) | Placebo Plus OBT (N=119)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 9 (10)
Lymphadenopathy (Blood and lymphatic system disorders) | 19 (24) | 4 (4)
Conjunctivitis (Eye disorders) | 17 (18) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 15 (18) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 25 (31) | 7 (8)
Abdominal pain upper (Gastrointestinal disorders) | 17 (19) | 11 (11)
Constipation (Gastrointestinal disorders) | 15 (19) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 75 (108) | 35 (41)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 7 (7)
Flatulence (Gastrointestinal disorders) | 17 (20) | 5 (7)
Haemorrhoids (Gastrointestinal disorders) | 8 (8) | 6 (6)
Nausea (Gastrointestinal disorders) | 41 (57) | 30 (40)
Vomiting (Gastrointestinal disorders) | 25 (41) | 17 (19)
Asthenia (General disorders) | 12 (13) | 2 (2)
Chest pain (General disorders) | 13 (15) | 4 (4)
Fatigue (General disorders) | 45 (57) | 18 (22)
Injection site reaction (General disorders) | 35 (41) | 14 (16)
Oedema peripheral (General disorders) | 12 (13) | 9 (10)
Pyrexia (General disorders) | 29 (32) | 24 (35)
Anogenital warts (Infections and infestations) | 12 (15) | 4 (4)
Bronchitis (Infections and infestations) | 34 (44) | 15 (18)
Cellulitis (Infections and infestations) | 11 (15) | 7 (7)
Folliculitis (Infections and infestations) | 12 (14) | 4 (4)
Furuncle (Infections and infestations) | 4 (4) | 6 (6)
Gastroenteritis (Infections and infestations) | 13 (14) | 6 (6)
Herpes zoster (Infections and infestations) | 27 (30) | 5 (5)
Influenza (Infections and infestations) | 17 (21) | 9 (14)
Nasopharyngitis (Infections and infestations) | 29 (50) | 15 (20)
Onychomycosis (Infections and infestations) | 8 (9) | 7 (8)
Oral candidiasis (Infections and infestations) | 12 (12) | 11 (12)
Pneumonia (Infections and infestations) | 14 (19) | 10 (14)
Sinusitis (Infections and infestations) | 35 (50) | 15 (18)
Upper respiratory tract infection (Infections and infestations) | 76 (114) | 29 (47)
Urinary tract infection (Infections and infestations) | 11 (12) | 11 (18)
Alanine aminotransferase increased (Investigations) | 18 (29) | 9 (11)
Aspartate aminotransferase increased (Investigations) | 20 (27) | 9 (12)
Blood bilirubin increased (Investigations) | 6 (7) | 6 (10)
Blood cholesterol increased (Investigations) | 10 (11) | 9 (11)
Blood creatine phosphokinase increased (Investigations) | 21 (24) | 8 (8)
Blood creatinine increased (Investigations) | 18 (37) | 11 (17)
Blood glucose increased (Investigations) | 13 (28) | 6 (7)
Blood phosphorus decreased (Investigations) | 3 (3) | 6 (8)
Blood triglycerides increased (Investigations) | 22 (30) | 14 (15)
Weight decreased (Investigations) | 14 (15) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 13 (16) | 10 (10)
Hyperlipidaemia (Metabolism and nutrition disorders) | 12 (12) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (32) | 15 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (27) | 14 (17)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 13 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (35) | 9 (12)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (23) | 8 (10)
Dizziness (Nervous system disorders) | 22 (27) | 10 (13)
Headache (Nervous system disorders) | 39 (62) | 19 (24)
Hypoaesthesia (Nervous system disorders) | 7 (10) | 8 (10)
Neuropathy peripheral (Nervous system disorders) | 15 (19) | 9 (11)
Paraesthesia (Nervous system disorders) | 10 (12) | 6 (7)
Anxiety (Psychiatric disorders) | 7 (7) | 13 (14)
Depression (Psychiatric disorders) | 15 (17) | 11 (12)
Insomnia (Psychiatric disorders) | 22 (27) | 11 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (32) | 21 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 7 (8)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (8)
Night sweats (Skin and subcutaneous tissue disorders) | 11 (15) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 30 (36) | 12 (17)
Hypertension (Vascular disorders) | 21 (21) | 5 (6)

LIMITATIONS AND CAVEATS:
Adverse events are reported by original treatment group for the entire 240-week study, including double-blind, open-label, and OLPVF phases; 83 of 119 participants in the placebo group also received raltegravir in the open-label or OLPVF phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial, but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.